CLINICAL TRIAL: NCT02537964
Title: Evaluation of the Effectiveness of Chlorhexidine Bathing in Reducing Nosocomial Infections in the Neonatal Intensive Care Unit
Brief Title: Effectiveness of Chlorhexidine Bathing in the Neonatal Intensive Care Unit
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: funding not available
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Maskit Bar-Meir, attending physician, Shaare Zedek Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 0018-15-SZMC
Record Dates: First submitted 2015-07-28; First posted 2015-09-02 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Infectious Disease Transmission
Keywords: chlorhexidine
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine bath (Experimental): Intervention: All infants in the NICU eligible for the study will be assigned for bathing three times a week with washcloths impregnated with 2% chlorhexidine gluconate
  Interventions: Other: washcloths impregnated with 2% chlorhexidine gluconate
- Standard bathing (No Intervention): Standard bathing with water +/- mild soap according to age and gestational week

INTERVENTIONS:
Other: washcloths impregnated with 2% chlorhexidine gluconate — All infants in the NICU eligible for the study will be assigned for bathing three times a week with washcloths impregnated with 2% chlorhexidine gluconate
  Other Names: Clinell ® Chlorhexidine wash cloths, GAMA healthcare
  Arms: Chlorhexidine bath

SUMMARY:
This is a prospective, controlled; crossover study of daily bathing with no-rinse, 2% chlorhexidine gluconate (CHG) impregnated washcloths versus bathing with water/soap or water according to gestational age and weight (e.g. standard bathing). The trial will take place in the Neonatal intensive care unit (NICU).

Baseline data ragarding bloodstream infections (BSI) and colonization with multidrug resistant orgnisms (MDRO) will be collected for 3-6 months prior to patient enrollment. In the preliminary phase of the study we will establish the safety of chlorhexidine bathing using Clinell ® Chlorhexidine wash cloths on three groups of patients: term infants admitted to the NICU; late preterm infants (34-37 weeks); preterm infants 30-34 weeks of gestation. Interim analysis for adverse events will be performed after each group of patients.

In the subsequent phases of the study, all infants admitted to the NICU and enrolled in the study will be bathed three times a week with Chlorhexidine wash cloths during the initial 6-months study period (intervention), followed by standard bathing during the second 6-months period, then again intervention period for 6 months and standard bathing for 6-months. Total study period- 3 years.

Data collection will include all bloodstream infections as well as surveillance cultures

DETAILED DESCRIPTION:
The study will take place in the Neonatal intensive care unit (NICU) of Shaare-Zedek Medical Center

Baseline data ragarding bloodstream infections (BSI) and colonization with multidrug resistant orgnisms (MDRO) will be collected for 3-6 months prior to patient enrollment.

Preliminary study:

In order to establish safety , we will enroll infants admitted to the NICU to three successive treatment groups , as follows: the first group will include term infants admitted to the NICU (gestational age 37+6 and >7 days old), the second group will include near-term infants (gestational age > 34+0 to 36+6 weeks and >7 days old) and the third group will include premature infants (gestational age >30+0 to 33+6 and >=10 days old). We intend to enroll up to 20 patients in each group, for a minimum of 200 patient days per group . All infants will be assigned for bathing three times a week with washcloths impregnated with 2% chlorhexidine gluconate (Clinell ® Chlorhexidine wash cloths, GAMA healthcare) for the duration of their NICU stay. The infant's skin will be monitored continuously as described below . In case of grade 3 or 4 reactions, the study interventions will be temporarily suspended, and the adverse event will be reported to the Helsinky committee and to the study steering committee. If no grade 3 or 4 reactions will be encountered after at least 200 patient days per group, enrollment to the subsequent group will be performed (e.g if no grade 3-4 reaction will be encountered for 200 patient days in group 1, we will start enrolling patients for group 2 etc.). If no grade 3-4 dermatitis is encountered in the preliminary study, we will initiate enrollment as described below.

In the subsequent phases of the study, :

All infants in the NICU eligible for the study will be assigned for bathing three times a week with washcloths impregnated with 2% chlorhexidine gluconate (Clinell ® Chlorhexidine wash cloths, GAMA healthcare) during the initial 6-months study period (intervention), followed by standard bathing during the second 6-months period, then again intervention period for 6 months and standard bathing for 6-months. Total study period- 2.5 years.

Inclusion criteria: infants weighing ≥1500 grams and >=10 days of age ; parents' informed consent Exclusion criteria: infants weighing <1500 grams or <10 days of age; parents' refusal to sign informed consent.

For standard bathing procedure see appendix 1.

Before the study initiation, as well as at the beginning of each study period, nurses will be instructed on the proper technique for bathing patients. Bathing will be performed according to product brochure, three times a week.

Outcome measures

A. Number of bacteremia episodes per 1000 patient days during the intervention periods compared with the control periods.

B. Number of new patients colonized with methicillin resistant Staphylococcus aureus (MRSA), vancomycin resitant enterococcus (VRE), carbapenem resistant Acinetobacter baumanii (CRAB) or extended spectrum beta-lactamase (ESBL) producing organisms per total number of patients, monthly range and variance.

C. Number of new patients colonized with MRSA, VRE, CRAB or ESBL per 1000 eligible patient days [ Total patient days - total patient days for patients identified with multidrug resistant organisms (MDRO)]

D. Time to colonization with MDRO during the intervention periods compared with the control periods.

Data collection:

Each patient admitted to the NICU during the study periods and meeting the inclusion criteria, will be recorded and assigned a specific study number. The dates of admission and dates of discharge will be recorded and used to calculate length of stay and to determine the incidence of nosocomial infections based on microbiological data. Clinical and laboratory data, including the use of invasive device (intravascular devices, mechanical ventilation, feeding tubes) will be collected on standardized forms. The data will be coded under a password protected database and linked only to study patient identifier.

Infections and MDRO acquisitions will be monitored during the study period. Events occurring within 2 days after the transition will be assigned to the previous bathing period.

For infection surveillance, daily review of cultures and new orders for antibiotic therapy will be performed for all study participants. Infectious events will be evaluated by an independent investigator blinded to the intervention period.

Active surveillance testing for MDRO will be performed once every two weeks during the study period. Swabs from the nasopharynx (for MRSA)] and from the rectal area (for ESBL producing organisms, VRE and CRAB) will be obtained by unit staff and processed in the microbiology laboratory of Shaare-Zedek Medical Center.

Trial oversight:

The steering committee of the study will include, except for the PI, an Infectious Disease physician and a neonatologist . There will be biweekly discussions of the progress report, reporting of compliance with active surveillance, reporting of compliance with bathing, and any adverse reactions or other problems.

Statistical analyses

Changes in the rates of BSI and clinical sepsis will be compared between the intervention and the control period. Continuous variables will be examined with the use of two-sample t-tests and linear regression modeling, and categorical variables will be examined by means of Fisher's exact test. Cox proportional-hazards regression model will be used to compare the time from admission until the first primary bloodstream infection , clinical sepsis or acquisition of MDRO between the control and intervention periods.

Sample size calculation: based on our ongoing surveillance, there are 2-3 BSI events per 1000 patients -days in our NICU. In order to detect a 50% reduction in BSI rates , the investigators will need 37,096 patient days (18,548 in each group) in order to have 80% power to reject the null hypothesis, with 0.05 level of significance. Currently, our average annual census is 45,000 patient days. therefore, a 2-year study will have >80% power to reject the null hypothesis (the BSI rates in the control period equal the rates in the intervention period).

Safety and monitoring.

A study that evaluated the tolerability of 2% CHG for catheter insertion antisepsis among infants ≥1500 grams and ≥7 days old found no significant dermatitis reactions . Seven of 48 infants had measurable CHG levels in the blood. In a trial that evaluated a multifactorial approach to reduce the rates of CLABSI, Andersen et al. noted that 4 of 36 neonates <1000g developed contact dermatitis after a 2% CHG scrub. There were no episodes of contact dermatitis in 49 study participants who were ≥1000g . The alternative for antisepsis in neonates is povidone-iodine. However, iodine absorption that may compromise thyroid function is one reason to explore the use of CHG. Although CHG was reported to be absorbed through neonatal skin in several trials, no significant systemic side effects were reported ' . Animal trials showed no significant toxicity from CHG . The US Food and Drug Administration (FDA) states on the drug facts box of 2% CHG cloth:" use with care in premature infants or infants under 2 months of age. These products may cause irritation or chemical burns".

Each participant's skin will be examined daily by nursing staff and twice a week by study personnel.

Skin reactions will be graded and recorded on a standard report form (appendix 2).

Grade 3 and 4 skin reactions will be reported as serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* infants weighing ≥1500 grams and >=10 days of age
* parents' informed consent

Exclusion Criteria:

* infants weighing <1500 grams or <10days of age;
* parents' refusal to sign informed consent.

Min Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09; Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
bacteremia episodes per 1000 patient days | 3 years
  Number of bacteremia events per 1000 patient days during the intervention periods compared with the control periods.

SECONDARY OUTCOMES:
Colonization with resistant bacteria | 2 years
  Number of new patients colonized with MRSA, VRE, CRAB or ESBL per total number of patients, monthly range and variance.
Time to colonization | 2 years
  Time to colonization with MDRO during the intervention periods compared with the control periods.
colonization with resistant bacteria | 2 years
  Number of new patients colonized with MRSA, VRE, CRAB or ESBL per 1000 eligible patient days [ Total patient days - total patient days for patients identified with MDRO]

CONTACTS AND LOCATIONS:
Overall Officials: Maskit Bar-Meir, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare-Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No